CLINICAL TRIAL: NCT00245674
Title: Solian Solution to Treat Schizophrenic Patients During an Acute Episode
Brief Title: SOLIACS: Solian Solution in the Acute Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM_L_0055; EudraCT # : 2004-004461-15
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Amisulpride

INTERVENTIONS:
Drug: amisulpride

SUMMARY:
During this study the efficacy and safety profile will be evaluated of the use of amisulpride in the form of a solution in schizophrenic patients with an acute episode.

The main purpose of the study is to observe the anti-psychotic effect of amisulpride as a solution during the first days of an acute episode of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenic in-patients with an acute episode
* aged between 18 and 65 years
* written informed consent

Exclusion Criteria:

* pregnancy and breast-feeding
* breast cancer, prolactinoma, pheochromocytoma
* hypersensitivity to amisulpride or one of the other excipients
* contra-indications when using amisulpride as per the SmPC

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-06

PRIMARY OUTCOMES:
*analyze the antipsychotic efficacy of amisulpride solution in the first days of an acute schizophrenic episode.

SECONDARY OUTCOMES:
*analyse the safety profile of amisulpride solution in treatment of schizophrenics with an an acute episode.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Christian Fassotte, M.D., Study Director — Sanofi
Locations (1):
- Sanofi-aventis, Diegem, Belgium